CLINICAL TRIAL: NCT02921347
Title: Efficacy and Safety of Switching Between Invasive and Noninvasive Ventilation to Facilitate Weaning in Difficult-weaning Patients: a Randomized Control Trial
Brief Title: Switching Between Invasive and Noninvasive Ventilation to Facilitate Weaning in Difficult-weaning Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, Principal Investigator, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cqykdxfsdyyy4
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Ventilator Weaning
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Patients in this group are received ventilator weaning by switching between invasive and noninvasive ventilation
  Interventions: Procedure: switching between invasive and noninvasive ventilation
- Control group (No Intervention): Patients in this group are weaned from ventilator as conventional methods.

INTERVENTIONS:
Procedure: switching between invasive and noninvasive ventilation — As defined criteria, patients are switched between invasive and noninvasive ventilation until the ventilator is successfully weaned.
  Arms: Intervention group

SUMMARY:
The aim of this study is to facilitate weaning by switching between invasive and noninvasive ventilation in difficult-weaning patients.

DETAILED DESCRIPTION:
This study only enrolled patients with tracheotomy. When a patient is eligible to this study, he or she is randomly assigned to intervention or control group.A patient in intervention group is switched to noninvasive ventilation by masking the tracheotomy tube. If the patient presents distress in noninvasive ventilation, he or she is switched to invasive ventilation. If the distress relieves, patient is switched to noninvasive ventilation again until the patient successfully weans from ventilator. In control group, the patient is weaned as the conventional methods.

ELIGIBILITY:
Inclusion Criteria:

* duration of invasive ventilation ≥14 days
* anticipation of difficult weaning
* Glasgow Coma Scale ≥13
* no upper airway obstruction
* presence of spontaneous breath

Exclusion Criteria:

* age less than 18 or more than 85 years
* contraindications for noninvasive ventilation
* anticipation of survival less than 6 months
* refusal of tracheotomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
ventilator weaning days | from enrollment to 90 days

SECONDARY OUTCOMES:
successful weaning rate | from enrollment to 90 days
ICU stay days | from admission to 90 days
hospital stay days | from admission to 90 days
ICU mortality | from admission to 90 days
hospital mortality | from admission to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Shuliang Guo, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The first affiated hospital, chongqing medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided